CLINICAL TRIAL: NCT00002546
Title: A Phase III Randomized Study of Accelerated Hyperfractionated Whole Abdominal Radiotherapy (AHWAR) Versus Combination Ifosfamide-Mesna With Cisplatin in Optimally Debulked Stage I, II, III, or IV Carcinosarcoma (CS) of The Uterus
Brief Title: Radiation Therapy Compared With Combination Chemotherapy in Treating Patients With Cancer of the Uterus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network)
Organization: GOG Foundation (Network)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: GOG-0150; CDR0000063303 (Other: NIH); ECOG-G150; NCI-2012-02226 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Sarcoma
Keywords: stage I uterine sarcoma; stage II uterine sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; uterine carcinosarcoma
MeSH Terms: conditions — Sarcoma | interventions — Cisplatin; Ifosfamide; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: ifosfamide
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether radiation therapy is more effective than combination chemotherapy in treating patients with cancer of the uterus.

PURPOSE: This randomized phase III trial is studying radiation therapy to see how well it works compared to combination chemotherapy in treating patients with cancer of the uterus.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the survival, progression-free interval, and failure patterns in patients with optimally debulked stage I-IV carcinosarcoma of the uterus treated with whole abdominal radiotherapy vs ifosfamide and cisplatin.
* Compare the incidence and type of acute and late adverse events observed with these treatment regimens in this patient population.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive whole abdominal radiotherapy 5 days a week for 4 weeks, followed by radiotherapy boost to the pelvis 5 days a week for 2.2 weeks.
* Arm II: Patients receive cisplatin IV followed by ifosfamide IV over 1 hour on days 1-4. Treatment continues every 3 weeks for 3 courses.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 216 patients will be accrued for this study within 6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary homologous or heterologous carcinosarcoma of the uterus (corpus and cervix)
* Surgical stage I-IV disease, including positive adnexa, tumor invading the serosa, positive pelvic and/or para-aortic nodes, involvement of the mucosa of the bowel, bladder, or rectum, intra-abdominal metastases, positive pelvic washings, or vaginal involvement within planned radiation port
* Prior total abdominal hysterectomy with bilateral salpingo-oophorectomy and maximum tumor resection of all gross intra-abdominal/pelvic disease, including grossly involved pelvic and para-aortic nodes within 8 weeks before study

  * No greater than 1 cm residual disease
* Cervical sarcomas also allowed
* No metastasis beyond the abdominal cavity at diagnosis, including the following:

  * Parenchymal liver metastasis
  * Lung metastasis
  * Positive inguinal lymph nodes
  * Positive scalene nodes
  * Radiographic or pathologic evidence of bone or brain metastasis

PATIENT CHARACTERISTICS:

Age:

* 21 and over

Performance status:

* GOG 0-2

Hematopoietic:

* WBC at least 3,000/mm3
* Granulocyte count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 1.5 times normal
* SGOT no greater than 3 times normal
* Albumin at least 3 g/dL
* No acute hepatitis

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 50 mL/min

Other:

* No septicemia
* No severe infection
* No severe gastrointestinal bleeding
* No prior invasive or concurrent malignancy within the past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Prior hormonal therapy allowed

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy

Surgery:

* See Disease Characteristics

Other:

* No prior therapy that would preclude study therapy

Ages: 21 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 1993-12; Primary Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron H. Wolfson, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center; Higinia R. Cardenes, MD, PhD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (65):
- United States (64):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Women's Cancer Center - Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Cancer Center, Orange, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Denver, Colorado
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - Hinsdale, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Cancer Center at Tufts - New England Medical Center, Boston, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler Air Force Base, Keesler Air Force Base, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at the Cooper University Hospital, Camden, New Jersey
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Gynecologic Oncology Network, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Abramson Cancer Center at the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Cancer Center at Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Southeast Gynecologic Oncology Associates, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Fletcher Allen Health Care - Medical Center Hospital of Vermont Campus, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Result] Wolfson AH, Brady MF, Rocereto T, Mannel RS, Lee YC, Futoran RJ, Cohn DE, Ioffe OB. A gynecologic oncology group randomized phase III trial of whole abdominal irradiation (WAI) vs. cisplatin-ifosfamide and mesna (CIM) as post-surgical therapy in stage I-IV carcinosarcoma (CS) of the uterus. Gynecol Oncol. 2007 Nov;107(2):177-85. doi: 10.1016/j.ygyno.2007.07.070. Epub 2007 Sep 5. PMID 17822748